CLINICAL TRIAL: NCT06719908
Title: A Double-blind, Placebo-controlled, Phase I Study of the Pharmacokinetic and Pharmacodynamic Interaction of Oral AFA-281 With Alcohol in Healthy Volunteers
Brief Title: A Phase I Study of the Interaction of Alcohol With Oral AFA-281 in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Afasci Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AFA-281-303
Record Dates: First submitted 2024-11-26; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Alcohol; Alcohol Use Disorders
Keywords: AFA-281; Alcohol; Ethanol; Healthy Volunteer
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AFA-281 with Ethanol (Active Comparator): AFA-281 (40 mg) will be administered as a single dose (oral) in combination with Alcohol (0.6 g/kg in females or 0.7g/kg in males).
  Interventions: Drug: AFA-281 is a small molecule, orally available; Other: Alcohol (Ethanol)
- AFA-281 with Ethanol Placebo (Placebo Comparator): AFA-281 (40 mg) will be administered as a single dose (oral) in combination with the Alcohol placebo (0.6 g/kg in females or 0.7g/kg in males).
  Interventions: Drug: AFA-281 is a small molecule, orally available
- AFA-281 placebo with Ethanol (Placebo Comparator): AFA-281 placebo (40 mg) will be administered as a single dose (oral) in combination with the Alcohol (0.6 g/kg in females or 0.7g/kg in males).
  Interventions: Other: Alcohol (Ethanol)
- AFA-281 placebo with Ethanol placebo (Sham Comparator): AFA-281 placebo (40 mg) will be administered as a single dose (oral) in combination with the Alcohol placebo (0.6 g/kg in females or 0.7g/kg in males).
  Interventions: Drug: AFA-281 is a small molecule, orally available; Other: Alcohol (Ethanol)

INTERVENTIONS:
Drug: AFA-281 is a small molecule, orally available — This is a study to evaluate the interaction of AFA-281 with alcohol
  Arms: AFA-281 placebo with Ethanol placebo; AFA-281 with Ethanol; AFA-281 with Ethanol Placebo
Other: Alcohol (Ethanol) — Alcohol will be administered in combination with AFA-281 or AFA-281 placebo
  Arms: AFA-281 placebo with Ethanol; AFA-281 placebo with Ethanol placebo; AFA-281 with Ethanol

SUMMARY:
The goal of this clinical trial is to evaluate if alcohol interacts with the drug candidate AFA-281 in adults (healthy volunteers). This trial will evaluate blood concentration levels of AFA-281 and ethanol. The main questions it aims to answer are: Does alcohol interact with AFA-281? What are the side effects (if any)? Researchers will compare AFA-281 to a placebo (a look-alike substance that contains no drug) to see if AFA-281 interacts with alcohol.

Participants will take a total of 4 treatment sessions separated by at least 2 days between treatments. The treatments will incorporate AFA-281 or placebo with ethanol or ethanol placebo. After each treatment vital signs will be monitored and blood collected to measure AFA-281 and ethanol levels. Participants will provide an assessment survey of symptoms. The total treatment time will be 9 inpatient days (8 nights), and a final follow-up visit 3 to 5 days after clinic discharge.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 4-way crossover study of the interaction of alcohol and oral AFA-281 in healthy adult volunteers. This study will evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) effects of co-administration of AFA-281 and ethanol in healthy, male and female subjects who are social or moderate drinkers but do not meet criteria for the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of Alcohol Use Disorder. Each subject will receive single doses of AFA-281, ethanol, placebo for AFA-481, and placebo for ethanol in a randomized, double-blind, crossover manner. Randomized blocks will be included to ensure that there is 1 day in between treatment sessions. Blood will be collected for PK and blood alcohol levels at pre-dose and at multiple timepoints after treatment. Safety parameters will be evaluated for tolerability such as vital signs and clinical pathology. Participants will provide an assessment survey of symptoms. The total treatment time will be 9 inpatient days (8 nights), and a final follow-up visit 3 to 5 days after clinic discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 21 and 55 years of age, inclusive.
* Must voluntarily sign and date each informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study specific procedures.
* Currently consumes alcohol regularly (defined as having consumed 7 to 21 standard drinks per week on average in the 6 months prior to screening and having consumed ≥5 standard drinks on at least one occasion in the 30 days prior to screening) but does not meet the DSM-5 criteria for Alcohol Use Disorder. Note: one standard alcoholic drink is equivalent to 1.5 oz. hard liquor or 5 oz. wine or 12 oz. beer.
* Body mass index (BMI) within the range of 18.5 to 30.0 kg/m2, inclusive.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG) at the screening visit
* Adequate venous access
* Must be surgically sterile (vasectomy, tubal ligation or hysterectomy) or agree to be sexually inactive or agree to use a barrier method of birth control (i.e., condom) from the start of screening until study completion, and agree to refrain from donating sperm, for 90 days after study drug administration.
* Agree to abstain from strenuous exercise during the inpatient stay of the study.

Exclusion Criteria:

* History of significant sensitivity to any drug.
* Has a clinically significant abnormal ECG or an ECG with a QTc interval corrected for heart rate using the Fridericia formula (QTcF) > 430 msec.
* Has an estimated creatinine clearance (CrCl) outside of normal range.
* History of head trauma with loss of consciousness, seizures or convulsions, including febrile, alcohol or drug withdrawal seizures.
* History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
* Requirement for any over-the-counter and/or prescription medication, vitamins and/or herbal supplements on a regular basis.
* Use of any medications, vitamins and/or herbal supplements within the 2-week period prior to study drug administration.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening and the results will be maintained confidentially by the study site.
* Display any latent signs of alcohol withdrawal per the Clinical Institute Withdrawal of Alcohol Assessment-Revised (CIWA-AR).
* History or current diagnosis of a substance use disorder.
* Positive urine drug screen for drugs of abuse at Screening or Day -1.
* Consumption of alcohol within the 1-day period prior to study drug administration.
* Receipt of any drug by injection within 30 days prior to study drug administration.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, endocrine, dermatological, metabolic or psychiatric disease or disorder, or any uncontrolled medical illness.
* A clinically notable vital sign abnormality including a history of syncopal or near syncopal events following abrupt change in posture.
* History of cardiac disease, including family history of long-QT syndrome, second degree heart block Type II, third degree heart block or unexplained sudden deaths in their family.
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration.
* Pregnant or nursing women
* Receipt of any investigational product within 6 weeks prior to study drug administration.
* Consumption of grapefruit or grapefruit products from 3 days prior to study drug administration.
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration.
* Current enrollment in another clinical study.
* Previous enrollment in this study.
* Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive AFA-281.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic evaluation of AFA-281 | Predose and 1, 2, 2.25, 2.5, 2.75, 3, 3.25, 4, 5, 6, 7, 8, 12 and 24 hours post dose
  Evaluation of AFA-281 concentrations in the blood over time
Evaluation of ethanol levels in the blood | Collected at 2, 2.25, 2.5, 2.75, 3, 3.25, 4, 5, 6, 7, 8, 12 and 24 hours post administration
  Measure ethanol concentrations in the blood over time
Dizziness visual analog scale (VAS) assessment | Collected at predose, 1, 2, 3, 4, 6 and 8 hours post dose
  Central nervous system test. Visual Analogue Scale for dizziness assessment on a scale 0 to 10. 0 no dizziness and 10 worst
Choice Reaction Time (CRT) evaluation | Predose and 1, 2, 3, 4, 6 and 8 hours post dose
  Central nervous system test. The subject is required to respond to one stimulus, the quicker the better
Balance Platform assessment | Predose and 1, 2, 3, 4, 6 and 8 hours post dose
  Central nervous system test. Balance platform assessment
Match to Sample Visual Search (MTS) assessments | 1, 2, 4 and 8 hours post dose
  Central nervous system test. Assesses attention and visual searching, with a speed accuracy trade-off. The quicker, the better.
Alertness visual analog scale (AVAS) | 1, 2, 4 and 8 hours post dose
  Central nervous system test. Asks a subject to indicate their feelings on a line with a scale from 0 mm on the left to 100 mm on the right. The scale can be used to assess sleepiness and other subjective experiences.

SECONDARY OUTCOMES:
Clinical chemistry | Baseline, pre-intervention and in 24 hours after completion of the intervention
  Blood test for metabolic panel
A complete blood count (CBC) with differential | Baseline, pre-intervention and in 24 hours after completion of the intervention
  complete blood count with differential
Heart Rate | Predose, 1, 2, 4 hours post dose
  Measurement of heart rate
Blood pressure, both systolic, and diastolic pressure | Predose, 1, 2, 4 hours post dose
  Measurement of blood pressure
Body weight | Baseline, pre-intervention and after in 24 hours of the intervention
  Measurement of body weight
Electrocardiogram (ECG) including P Wave, QRS Complex, and QT Interval, etc.) | Baseline, pre-intervention and 2 hours post dose
  ECG assessment

IPD SHARING:
Plan to Share IPD: Undecided